CLINICAL TRIAL: NCT02203448
Title: A Multi-centre, Prospective, Single-arm Post Market Clinical Follow up Study (PMCF) of the FACET WEDGE Spinal System to Assess Outcomes in Subjects With Chronic Low Back Pain Due to Degenerative Disc Disease (DDD), Facet Joint Disease and/or Pseudo Arthrosis Post Anterior Instrumentation
Brief Title: Facet Wedge Post Market Study
Status: Completed | Type: Observational
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CT13/01
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Chronic Low Back Pain; Degenerative Disc Disease; Facet Joint Disease; Pseudo Arthrosis Post Anterior Instrumentation
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FACET WEDGE spinal system: The FACET WEDGE spinal system provides additional stability to a spinal segment to enhance fusion conditions.
  Interventions: Device: Facet Wedge spinal system

INTERVENTIONS:
Device: Facet Wedge spinal system

SUMMARY:
A Multi-centre, Prospective, single-arm post market clinical follow up study (PMCF) of the FACET WEDGETM spinal system to assess outcomes in subjects with chronic low back pain due to Degenerative Disc Disease (DDD), facet joint disease and/or pseudo arthrosis post anterior instrumentation. The objective of this study is to assess outcomes following implantation of the FACET WEDGE spinal system when used to provide fixation of lumbar motion segments.

The primary objective of this study is to determine the rate of re-operations at the index level(s).

The secondary objectives of this study are to confirm the safety and performance of the device and to collect patient reported outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with at least one of the following:

   * Degenerative Disc Disease (DDD);
   * Degenerative facet joint disease (isolated facet based symptomatic back pain);
   * Pseudoarthrosis post anterior instrumentation;
2. Subjects who are a fusion candidate for single or multiple levels fusion between L1-S1;
3. Subjects, who, in the opinion of the Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

Exclusion Criteria:

Preoperative exclusion criteria:

1. Segmental instability of the index level in case of planned stand-alone FACET WEDGE usage;
2. Unilateral application , except in combination with pediclescrew fixation on the contralateral side;
3. Compromised facets due to decompression techniques;
4. Spondylolisthesis;
5. Fracture or other instabilities of the posterior elements;
6. Tumor;
7. Acute or chronic systemic or localized spinal infections;
8. Nursing mothers or women who are pregnant or plan to become pregnant during the time of the study;
9. Subjects aged below 18 years;
10. Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation;

    Intraoperative exclusion criteria:
11. Intraoperative decision to use implants other than the device under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cases in the cohort are selected from patients treated in hospitals.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
reoperation rate at the index level(s) | at two years

SECONDARY OUTCOMES:
the radiographic range of motion (ROM) at the index levels | Pre-treatment, 6 months, 12 months, 24 months
patient (back and leg) pain reported on a Numeric Rating Scale (NRS) | pre-treatment, prior to D/C, 6 weeks, 6 months, 12 months, 24 months.
functional success based on results from the Oswestry Disability Index (ODI) | Pre-treatment, 6 weeks, 6 months, 12 months, 24 months
Adverse events | Throughout the study
  The nature and incidence of all procedural and post-treatment adverse events will be recorded and reported appropriately throughout the study to assess safety.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kandziora, PhD, Principal Investigator — Berufsgenossenschaftliche Unfallklinik, Frankfurt am Main, Germany
Locations (3):
- Germany (2):
  - BG Unfallklinik, Frankfurt am Main
  - Schon Klinik Munchen, München
- UVN, Ružomberok, Slovakia